CLINICAL TRIAL: NCT04171453
Title: POST-MARKETING SURVEILLANCE (PMS) TO OBSERVE THE SAFETY AND EFFECTIVENESS OF LYRICA(REGISTERED) CR EXTENDED RELEASE TABLETS
Brief Title: Post-marketing Surveillance (PMS) to Observe the Safety and Effectiveness of Lyrica CR Extended Release Tablets
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Viatris Korea (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: A0081364
Record Dates: First submitted 2019-10-10; First posted 2019-11-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open-label: This study was open-label with only one treatment group. Lyrica CR was prescribed in accordance with usual clinical practice.
  Interventions: Drug: Lyrica CR (Pregabalin)

INTERVENTIONS:
Drug: Lyrica CR (Pregabalin) — Lyrica CR 82.5mg, 165mg, or 330mg OD

SUMMARY:
This is an open-label, non-comparative, non-interventional, prospective, and multi-center PMS study to observe safety and effectiveness of Lyrica CR (82.5mg, 165mg, 330mg) in Korean subjects under the actual condition of use. PMS is an obligation to K-MFDS.

ELIGIBILITY:
[Inclusion criteria]

To be eligible to enter this study, the subject will have to meet the following inclusion criteria:

1. Korean patients who have been administered Lyrica CR for the first time according to the current local labeling (indication, dosage and administration).
2. Subjects who have consented to participate in this study by signing the data privacy statement.

[Exclusion criteria]

Patients meeting any of the following criteria will not be included in the study:

1. Patients who have deviated from local labeling (indication, dosage and administration) in taking this drug
2. Renal impairment patients with CLCr less than 30 mL/min or who are undergoing hemodialysis.
3. Patients who have hypersensitivity to the active substance (pregabalin) or to any of the excipients.
4. Other patients who are decided to be not prescribed by the investigator under the routine medical practice, considering the balance the overall risk and benefit, for example, patients have suicidal behavior and ideation, or have any risk of these, and/or patients who are in pregnancy or lactation, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects administered with Lyrica CR as a part of routine treatment who comply with the local labeling.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-07-14 (Estimated); Study Completion 2022-07-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Event (AE) | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  Duration, severity, outcome and causal relationship of the AE with the study drug (Lyrica CR) will be measured.
Number of participants with Adverse Drug Reactions (ADRs) | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  All the AEs, except for those with the causal relationship of 'Unlikely', are considered as adverse drug reactions (ADRs)
Number of participants with Serious Adverse Event (SAE) | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  SAE is any untoward medical occurrence attributed to Lyrica CR in a participant who received the study drug. A serious ADR was an ADR resulting in any of the following outcomes or deemed signification for any other reason: death; life-threatening; requires inpatient hospitalization or prolongation of hospitalization; results in persistent or significant disability/incapacity; results in congenital anomaly/birth defects; is an important medical event.
Number of participants with unexpected AEs | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  Unexpected AEs will be classified by medical review with reference to the local product document. Events already included in the "Precautions for use" section of the local product document will be classified as "expected". All other events that are not included in the "Precautions for use" section of the local product document will be classified as "unexpected".
Number of participants with unexpected ADRs | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  Unexpected ADRs will be classified by medical review with reference to the local product document. Events already included in the "Precautions for use" section of the local product document will be classified as "expected". All other events that are not included in the "Precautions for use" section of the local product document will be classified as "unexpected".
Percentage of participants with Adverse Event (AE) | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  Duration, severity, outcome and causal relationship of the AE with the study drug (Lyrica CR) will be measured.
Percentage of participants with Serious Adverse Event (SAE) | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  SAE is any untoward medical occurrence attributed to Lyrica CR in a participant who received the study drug. A serious ADR was an ADR resulting in any of the following outcomes or deemed signification for any other reason: death; life-threatening; requires inpatient hospitalization or prolongation of hospitalization; results in persistent or significant disability/incapacity; results in congenital anomaly/birth defects; is an important medical event.
Percentage of participants with Adverse Drug Reactions (ADRs) | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  All the AEs, except for those with the causal relationship of 'Unlikely', are considered as adverse drug reactions (ADRs)
Percentage of participants with unexpected AEs | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  Unexpected AEs will be classified by medical review with reference to the local product document. Events already included in the "Precautions for use" section of the local product document will be classified as "expected". All other events that are not included in the "Precautions for use" section of the local product document will be classified as "unexpected".
Percentage of participants with unexpected ADRs | Maximum of 12 weeks (window period of 2 weeks) from the time of initial administration of Lyrica CR.
  Unexpected ADRs will be classified by medical review with reference to the local product document. Events already included in the "Precautions for use" section of the local product document will be classified as "expected". All other events that are not included in the "Precautions for use" section of the local product document will be classified as "unexpected".

SECONDARY OUTCOMES:
Severity of pain after administration of Lyrica CR | At 12 weeks (window period of 2 weeks) or at the time of drug discontinuation.
  The severity of pain will be recorded by daily average pain score in 24 hours recall period, calculated with 11-point Numeric Rating Scale (NRS).
Sleep interference status after administration of Lyrica CR | At 12 weeks (window period of 2 weeks) or at the time of drug discontinuation.
  The sleep interference status is recorded by the answer with 11-point Likert scale (0=did not interfere, 10=unable to sleep) from the question, "How much did the pain interfere with your sleep during the past 24 hours?" and the data will be based on the patient's recall
Patient's Global Impression of Change (PGIC) | At the end of the study (At 12 weeks, with window period of 2 weeks)
  Rating is given by the subject to indicate the impression of change since baseline. This rating is on a 7-point scale that has categories such as 'very much improved', 'much improved', 'a little improved', 'no change', 'a little worse', 'much worse', and 'very much worse'.
Clinician's Global Impression of Change | At the end of the study (At 12 weeks, with window period of 2 weeks)
  Rating is given by the investigator to indicate the impression of change since baseline based on the Severity of pain after administration, the Sleep interference status after administration, and the PGIC. This rating is on a 7-point scale that has categories such as 'very much improved', 'much improved', 'a little improved', 'no change', 'a little worse', 'much worse', and 'very much worse'.
Final Effectiveness Evaluation | At the end of the study (At 12 weeks, with window period of 2 weeks)
  On the results of the above Clinician's Global Impression of Change, the investigator shall mark 'very much improved', 'much improved', and 'a little improved' as 'valid', or mark 'no change', 'a little worse', 'much worse', and 'very much worse' as 'invalid'.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Gyeongsang National University Changwon Hospital, Changwon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Hospital Clinical Research Institute, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A0081364